CLINICAL TRIAL: NCT06603584
Title: Phenotypes of Preschool Wheezing Among Children Attending Sohag University Hospital
Status: Recruiting | Type: Observational
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Amr Ahmed Gamal Eldin, Resident-pediatric department-sohag hospital university, Sohag University
Other Study IDs: soh-Med-24-06-20MS
Record Dates: First submitted 2024-09-17; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Wheezing
MeSH Terms: conditions — Respiratory Sounds | interventions — X-Rays

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- group A: Bronchial Asthma
  Interventions: Radiation: Chest x- Rays
- group B: Chronic Aspiration
  Interventions: Radiation: Chest x- Rays
- group C: Primary Ciliary Dyskinesia
  Interventions: Radiation: Chest x- Rays
- group D: Cystic Fibrosis
  Interventions: Radiation: Chest x- Rays

INTERVENTIONS:
Radiation: Chest x- Rays — prebronchial Thicknening - Right upper lobe Patches suggesting Aspiration -Collapsing lobe

SUMMARY:
Wheezing in preschool children is very common, with a wide differential diagnosis. It is essential to be sure of the exact sound that parents are describing; the term 'wheeze' is often applied to non-specific sound.Approximately one-third of children are diagnosed with wheeze in the first 3 years of life, making wheeze one of the commonest respiratory symptoms.The differential diagnosis of wheeze is wide, and different management strategies are needed depending on the underlying phenotype. The word 'wheeze' is used to describe many different sounds. That can be heard by both clincians and parent. Even if true wheeze is heard, this should not be automatically assumed to be due to bronchospasm. Airway narrowing by mucus will produce true wheeze but does not respond to bronchodilators. Similarly, airway malacia, either related to intrinsic airway wall defects or loss of alveolar tethering points, are also causes of bronchodilatorunresponsive wheeze; indeed, bronchodilators, by reducing airway smooth muscle tone, may actually worsen airway narrowing.

ELIGIBILITY:
Inclusion Criteria:

* patients from the age of one to five years with recurrent wheezing

Exclusion Criteria:

* Children above 5 years and below one year old.
* Failure to obtain informed consent.
* Children below 6 years with chest diseases other than wheezing

Ages: 2 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: - patients from the age of one to five years with recurrent wheezing
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-06-04 (Actual); Primary Completion 2025-04-04 (Estimated); Study Completion 2025-04-04 (Estimated)

PRIMARY OUTCOMES:
Forced Expiratory Volume | 6 months
  Changes in Forced Expiratory Volume in bronchial Asthmatic Patient

CONTACTS AND LOCATIONS:
Locations (1):
- Sohag university Hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Fitzpatrick AM, Bacharier LB, Guilbert TW, Jackson DJ, Szefler SJ, Beigelman A, Cabana MD, Covar R, Holguin F, Lemanske RF Jr, Martinez FD, Morgan W, Phipatanakul W, Pongracic JA, Zeiger RS, Mauger DT; NIH/NHLBI AsthmaNet. Phenotypes of Recurrent Wheezing in Preschool Children: Identification by Latent Class Analysis and Utility in Prediction of Future Exacerbation. J Allergy Clin Immunol Pract. 2019 Mar;7(3):915-924.e7. doi: 10.1016/j.jaip.2018.09.016. Epub 2018 Sep 26. PMID 30267890
- [Background] Lowe LA, Simpson A, Woodcock A, Morris J, Murray CS, Custovic A; NAC Manchester Asthma and Allergy Study Group. Wheeze phenotypes and lung function in preschool children. Am J Respir Crit Care Med. 2005 Feb 1;171(3):231-7. doi: 10.1164/rccm.200406-695OC. Epub 2004 Oct 22. PMID 15502115
- [Background] Salehian S, Fleming L, Saglani S, Custovic A. Phenotype and endotype based treatment of preschool wheeze. Expert Rev Respir Med. 2023 Jul-Dec;17(10):853-864. doi: 10.1080/17476348.2023.2271832. Epub 2023 Nov 24. PMID 37873657
- [Background] Kwong CG, Bacharier LB. Phenotypes of wheezing and asthma in preschool children. Curr Opin Allergy Clin Immunol. 2019 Apr;19(2):148-153. doi: 10.1097/ACI.0000000000000516. PMID 30640211